CLINICAL TRIAL: NCT03928756
Title: Adaptive Interventions for Prevention/Intervention for Youth Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Maureen A Walton, Professor of Psychiatry, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00148393
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Substance Use
Keywords: substance use; mobile health
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-participant randomization (Experimental): Each day, each available participant will be randomly assigned to receive either: a push notification with tailored intervention content; a push notification with engaging, nontherapeutic content; or no push notification.
  Interventions: Behavioral: Push Notifications with Tailored Intervention Content; Behavioral: Push Notifications with Engaging, Non-therapeutic Content; Behavioral: No Push Notifications

INTERVENTIONS:
Behavioral: Push Notifications with Tailored Intervention Content — Participants will receive a push notification with a therapeutic message (e.g., about stress, mood, substance use motives, tools to reduce risky substance use) tailored to their recent daily or weekly survey responses. Messages include visual (memes, images, videos) and written content.
Behavioral: Push Notifications with Engaging, Non-therapeutic Content — Participants will receive a push notification with an engaging, non-therapeutic message (e.g., fun facts).
Behavioral: No Push Notifications — Participants will not receive a push notification.

SUMMARY:
The main aim of this formative study is to test and iteratively refine a new mobile phone app, which delivers assessments and tailored intervention content. The study will use social media advertisements to recruit a total of 40 youth between the ages of 16-24 years. Those screening positive for past-month binge drinking or marijuana use will be invited to complete a baseline survey, download and use the app for 30 days, and complete a follow-up survey about the app functionality, design and content, and preliminary outcomes (intentions and importance of reducing use).

DETAILED DESCRIPTION:
Previously, the study team developed a prototype mobile application which utilized novel engagement strategies to enhance user adherence with daily and weekly survey assessments. The new app developed for this study extends the previous app by featuring the capability to also deliver tailored health intervention. As part of the app, users are prompted to complete brief daily and weekly assessments for 30 days. For each completed assessment, users earn small financial rewards and points to unlock new fish that populate a virtual aquarium in the app. The app also features push notifications with survey reminders and life insights (or graphs plotting data collected over time) to increase user engagement with the app. Additionally, each day, users are randomized to receive intervention content (see the "Interventions" section for more information) tailored on their recent assessment responses. After 30 days of using the app, participants will be asked to complete a follow-up survey; data collected will provide preliminary feedback regarding the feasibility and effectiveness of using the app to deliver substance use intervention content to affected youth.

ELIGIBILITY:
Inclusion Criteria:

1. Have an iPhone smartphone on which the app can be downloaded
2. Self-reported past-month binge drinking (4/5 or more drinks on one occasion, tailored by sex) OR any past-month marijuana use without a medical marijuana card
3. Meet study verification criteria (i.e., use of CAPTCHA, IP address checks, social media checks).

Exclusion Criteria:

1. Unable to understand English

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Change in Intentions to Reduce Alcohol Use | 1-month post-app start
  Change in intentions to reduce alcohol use will be assessed using a 10-point validated Likert item which asks participants to rate their current likelihood of cutting back on their alcohol use. (a score of 1 is equivalent to not at all likely and a score of 10 is very likely)
Change in Importance of Reducing Alcohol Use | 1-month post-app start
  Change in importance of reducing alcohol use will be assessed using a 10-point validated Likert item which asks participants to rate how important it is to them to cut back on their alcohol use. (a score of 1 is equivalent to not at all important and a score of 10 is very important)
Change in Intentions to Reduce Marijuana Use | 1-month post-app start
  Change in intentions to reduce marijuana use will be assessed using a 10-point validated Likert item which asks participants to rate their current likelihood of cutting back on their marijuana use. (a score of 1 is equivalent to not at all likely and a score of 10 is very likely)
Change in Importance of Reducing Marijuana Use | 1-month post-app start
  Change in importance of reducing alcohol use will be assessed using a 10-point validated Likert item which asks participants to rate how important it is to them to cut back on their marijuana use. (a score of 1 is equivalent to not at all important and a score of 10 is very important)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen Walton, MPH, PHD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-06-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03928756/ICF_000.pdf